CLINICAL TRIAL: NCT00301652
Title: Mycophenolate Mofetil Versus Cyclophosphamide in the Induction Treatment of ANCA Associated Vasculitis
Brief Title: MMF Versus CTX in the Induction Treatment of ANCA Associated Vasculitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nanjing University School of Medicine (Other)
Responsible Party: Research Institute of Nephrology, Jinling Hospital, Nanjing University School of Medicine, Nanjing University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NJCT-0607
Record Dates: First submitted 2006-03-10; First posted 2006-03-13 (Estimated); Last update posted 2010-06-08 (Estimated); Status verified 2009-03

CONDITIONS: Vasculitis; Anti-Neutrophil Cytoplasmic Antibody
Keywords: ANCA; vasculitis; mycophenolate mofetil; cyclophosphamide; treatment
MeSH Terms: conditions — Vasculitis | interventions — Mycophenolic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- mycophenolate mofetil (Experimental)
  Interventions: Drug: mycophenolate mofetil

INTERVENTIONS:
Drug: mycophenolate mofetil — MMF,1.0g/d
  Other Names: MMF,cellcept,mycophenolate mofetil

SUMMARY:
The purpose of this study is to access the efficacy of MMF compared to CTX in inducing remission and improving renal function in subjects with ANCA associated vasculitis with renal involvement.

DETAILED DESCRIPTION:
The ANCA-associated vasculitides can be life threatening. Glucocorticoids and cyclophosphamide therapy is effective in about 80% patients. However, the side effects such as bone marrow suppression, infection, cystitis, infertility, myelodysplasia preclude further use of cyclophosphamide in some patients and the relapse rate is high.

Recent studies have shown that mycophenolic acid(MPA), the active metabolite of mycophenolate mofetil(MMF), could exhibit multifarious effects on endothelial cells, including inhibition of ICAM-1 expression, neutrophil attachment,IL-6 secretion, and the process of angiogenesis, which contribute to the efficacy of MMF in the treatment of vasculitic lesions such as lupus nephritis with vasculitic lesions. This study was a feasibility study to assess the safety and effectiveness of MMF in inducing remission in subjects with ANCA-associated SVV compared with pulse intravenous cyclophosphamide. After enrollment, subjects were followed longitudinally, and formal measurements of disease activity were determined using the Birmingham Vasculitis Activity Score (BVAS).

ELIGIBILITY:
Inclusion Criteria:

1. A new diagnosis of ANCA associated vasculitis (eg. MPA or Wegener granulomatous, or renal limited vasculitis) proved by histology and serology.
2. Renal involvement attributable to active ANCA associated vasculitis with at least one of the following:

   * Elevated serum creatinine between 150 and 500 umol/l - renal biopsy
   * Demonstrating paucin -immune necrotizing glomerulonephritis
   * Red cell casts
   * Haematuria with > 30 red blood cells/HPF and proteinuria > 1g/24h
3. Serum ANCA positive by indirect immunofluorescence (IIF) and positivity in the anti-PR3 or anti-MPO by ELISA
4. Age 18~65 years

Exclusion Criteria:

1. More than two weeks treatment with cyclophosphamide (CYC) or other cytotoxic drug within previous 6 months or with oral corticosteroids (OCS) for more than 4 weeks
2. Co-existence of another multisystem autoimmune disease, e.g. SLE
3. Serum creatinine > 500umol/l
4. Severe viral infection(HBV, HCV, CMV) within 3 months of first randomization or known HIV infection
5. Congenial or acquired immunodeficiency
6. Immediately life-threatening organ manifestations (e.g. lung haemorrhage or dialysis dependence)
7. Previous malignancy
8. Pregnancy or inadequate contraception if female
9. Anti-GBM antibody positivity
10. Cerebral infarction due to vasculitis
11. Rapidly progressive optic neuropathy or retinal vasculitis or orbital pseudotumour
12. Massive gastro-intestinal bleeding
13. Heart failure due to pericarditis or myocarditis
14. Liver dysfunction measured on at least 2 separate occasions
15. Age < 18y or Age > 65y

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2003-06; Primary Completion 2004-04 (Actual); Study Completion 2005-12 (Actual)

PRIMARY OUTCOMES:
The efficacy of MMF compared to CTX in inducing remission and improving renal function in subjects with ANCA associated vasculitis. | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Lei-Shi Li, M.D., Study Chair — Research Institute of Nephrology, Jinling Hospital, Nanjing University School of Medicine
Locations (1):
- Research Institute of Nephrology, Jinling Hospital, Nanjing University School of Medicine, Nanjing, Jiangsu, China